CLINICAL TRIAL: NCT07218965
Title: Fostering Agricultural Relationships and Meaning - Thriving on Kinship (FARM-TOK)
Brief Title: Fostering Agricultural Relationships and Meaning - Thriving on Kinship
Acronym: (FARM-TOK)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20250176
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Loneliness; Social Isolation; Rural Health
MeSH Terms: conditions — Social Isolation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental): CBT delivered over the course of 6, ~45 minute sessions delivered via telehealth
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Perceived Social Isolation
- Therapist-delivered Health Education (Active Comparator): Health education sessions delivered over the course of 6, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Perceived Social Isolation — Consists of six sessions focused on addressing thoughts, emotions, and behaviors that maintain feeling alone as a way to reduce loneliness and substance use.
  Other Names: CBT-PSI
  Arms: Cognitive-Behavioral Therapy
Behavioral: Health Education — Health education provides information on the importance and benefits of and guidelines for living a health lifestyle.
  Other Names: HET
  Arms: Therapist-delivered Health Education

SUMMARY:
This study aims to enroll 65 participants who will be assigned to one of two groups. Each group will receive an intervention consisting of six weekly sessions of 40-60 minutes each. Eligibility includes residing in an agricultural area and reporting loneliness or feeling alone or disconnected.

DETAILED DESCRIPTION:
Individuals (n = 65) who reside in a agricultural area and report loneliness will be randomized to either (1) therapist-delivered cognitive-behavioral therapy for perceived social isolation, or (2) therapist-delivered Health Education. Loneliness, quantity of social interactions, perceived social support, substance use outcomes, and other key outcomes and descriptive characteristics will be assessed at baseline, mid-treatment, post-treatment, and at a one-month follow-up. Participants will have the option to complete daily ecological momentary assessments (EMA) 3 times a day for 7 weeks via an app on their smartphone, Catalyst by MetricWire, throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to provide informed consent
* understand English
* have internet access
* reside in an agricultural area
* screen positive for loneliness by scoring at least 44 on the 20-item UCLA Loneliness Scale

Exclusion Criteria:

* unable to give informed consent
* non-English speaking
* does not have consistent access to a phone and/or internet
* reports being diagnosed with a neurological disorder or a current psychotic or bipolar 1 diagnosis
* current suicidal or homicidal intent indicating a need for immediate hospitalization or treatment as determined by clinical interviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in loneliness | Baseline to 6 months
  Loneliness will be measured using the UCLA Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
Mean change in anxiety | Baseline to 6 months
  Anxiety will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Mean change in depression | Baseline to 6 months
  Depression will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Mean change in social interactions | Baseline to 6 months
  Duke Social Support Index assesses several domains of perceived social support, including social network size, social interaction, social satisfaction, and instrumental social support. Higher scores indicate a higher quality of social interactions. Scores range from 0 to 37.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Department of Psychiatry and Behavioral Health, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified demographic and clinical data collected as part of this project will be available as raw individual level data for sharing with external researchers working at an institution with a Federalwide Assurance (FWA) for the Protection of Human Subjects. Data will therefore be available for secondary analytic purposes. Names and institutions of persons either given or denied access to data will be tracked by our Administrative Core and will be available upon request from the sponsor. Data will not be available for data sharing until after this project is complete and the primary outcomes are published.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for at least the next two years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).